CLINICAL TRIAL: NCT01826812
Title: Functional Impairment of Reading Ability in Dry Eye Patients and Effects of Sustained Reading on the Ocular Surface
Brief Title: Impairment of Reading Ability in Dry Eye Patients
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: NA_00082755
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2017-08

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tears
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dry Eye: The patients with Sjogren Syndrome related or non-Sjogren Syndrome related dry eye. The participants will be asked some questions. Before and after reading a text silently in 30 minutes "30 minutes sustained reading", a detailed dry eye exam will be performed.
  Interventions: Other: 30 minutes sustained reading; Other: Dry eye exam
- Controls: The patients without dry eye. The participants will be asked some questions. Before and after reading a text silently in 30 minutes "30 minutes sustained reading", a detailed dry eye exam will be performed.
  Interventions: Other: 30 minutes sustained reading; Other: Dry eye exam

INTERVENTIONS:
Other: 30 minutes sustained reading — The participants will be given a text to read silently in 30 minutes.
Other: Dry eye exam — Tear break-up time, tear collection, osmolarity, Schirmer test, corneal and conjunctival staining.

SUMMARY:
To assess the reading function impairment in patients with dry eye and to assess the effects of reading on the ocular surface.

DETAILED DESCRIPTION:
This study is being done to understand how reading is affected in people with dry eye in comparison with healthy controls and what effect reading has on the ocular surface in patients with dry eye.

ELIGIBILITY:
Inclusion Criteria:

* age of 50 or greater,
* literacy in English language,
* ability to give informed consent

Exclusion Criteria:

* binocular vision below 20/25,
* any ocular surgery within the last 3 months,
* mental issues,
* illiteracy,
* language problems which might possibly interfere with reading ability,
* history of taking or current use of topical prescription anti-inflammatory eye drops (including, cyclosporine and steroids as well as any glaucoma eye drops).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with known dry eye as well as normal healthy control subjects with no ocular surface diseases will be recruited from the Ocular Surface Diseases and Dry Eye Clinic as well as Glaucoma Clinic of the Wilmer Eye Institute.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esen K Akpek, MD, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Wilmer Eye Institute, Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ocular staining score (OSS) is sum of the corneal and conjuctival staining scores with a total possible maximum score of 12 for each eye. Corneal staining is graded with a maximum possible fluorescein score of 6 for each eye. Nasal and temporal conjunctiva are graded separately with a lissamine green staining score between 0 and 3 for each area.
Groups:
- Dry Eye: Dry eye defined as OSDI score more than 12 and/or total OSS score 3 and more
- Controls: Controls defined as OSDI 12 and less AND total OSS score less than 3
Period: Overall Study
Arm/Group | Dry Eye | Controls
Started | 167 | 33
Completed | 167 | 32
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dry Eye | Controls | Total
Number analyzed (Participants) | 167 | 33 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.7) | 61.4 (8.7) | 63.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 19 | 141
  Male | 45 | 14 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 160 | 32 | 192
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 6 | 23
  White | 139 | 24 | 163
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 167 | 33 | 200
Baseline Visual Acuity, logMAR [Mean (Standard Deviation); unit: logMAR] | -0.04 (0.11) | -0.03 (0.10) | -0.038 (0.11)
Baseline Osmolarity [Mean (Standard Deviation); unit: mOsm/L] | 312 (28) | 306 (10) | 311 (26)
Baseline total OSS score [Mean (Standard Deviation); unit: scores on a scale of 0 to 12] — Ocular staining score (OSS) is sum of the corneal and conjuctival staining scores with a total possible maximum score of 12 for each eye. Corneal staining is graded with a maximum possible fluorescein score of 6 for each eye (the punctate epithelial erosions grade between 0-3 plus any extra points for modifiers up to 3). Nasal and temporal conjunctiva are graded separately with a score range between 0 and 3 for each area after instillation of lissamine green. An abnormal OSS is defined as being a total score of 3 or more.
  scores on a scale of 0 to 12 | 4.9 (3.3) | 0.9 (0.9) | 4.3 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Sustained Silent Reading Speed
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: words/minute
Arm/Group | Dry Eye | Controls
Number analyzed (Participants) | 167 | 32
words/minute | 248.4 (79.5) | 270.3 (75.3)

2. Secondary Outcome: Change in Total Ocular Staining Score (OSS)
Description: Ocular staining score (OSS) is sum of the corneal and conjuctival staining scores with a total possible maximum score of 12 for each eye. Corneal staining is graded with a maximum possible fluorescein score of 6 for each cornea (the punctate epithelial erosions grade between 0-3 plus any extra points for modifiers up to 3). Nasal and temporal conjunctiva are graded separately with a score range between 0 and 3 for each area after instillation of lissamine green. An abnormal OSS is defined as being a total score of 3 or more.
Time Frame: Before and after 30 minutes reading
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dry Eye | Controls
Number analyzed (Participants) | 167 | 32
units on a scale | 1.5 (1.4) | 1.1 (1.2)

3. Secondary Outcome: Change in Tear Osmolarity
Time Frame: Before and after 30 minutes reading
Measure: Mean (Standard Deviation); unit: mOsm/L
Arm/Group | Dry Eye | Controls
Number analyzed (Participants) | 167 | 32
mOsm/L | 2.7 (12.3) | 1.8 (10.9)

4. Secondary Outcome: Change in Visual Acuity
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Dry Eye | Controls
Number analyzed (Participants) | 167 | 32
logMAR | 0.02 (0.07) | 0.02 (0.09)

5. Secondary Outcome: Cytokines
Description: Identification of various inflammatory cytokines in tear film of dry eye patients comparing to controls.
Time Frame: Tear samples were collected on the day of the exam. The samples were frozen to be assayed upon completion of the study.
Population: The cytokine analysis was performed in the samples of selected participants based on their clinical signs and characteristics. The sample size of the groups was justified using the power analysis.
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Dry Eye: Patients with Sjogren Syndrome related or non-Sjogren Syndrome related dry eye.
- Controls: Participants without dry eye.
Arm/Group | Dry Eye | Controls
Number analyzed (Participants) | 42 | 21
pg/mL
  IFNg | 99.79 (16.81) | 150.10 (30.29)
  TNFa | 131.16 (54.63) | 107.53 (25.30)
  IL6 | 130.78 (39.65) | 69.64 (13.40)
  IL17A | 176.08 (28.39) | 200.00 (41.42)
  IL1b | 27.40 (5.09) | 27.87 (6.47)
  IL8 | 903.91 (268.02) | 157.58 (32.39)
  IL10 | 211.69 (30.37) | 304.29 (55.01)
  IL12p70 | 70.89 (10.06) | 131.32 (28.59)

ADVERSE EVENTS:
Time Frame: Started with the first patient enrollment on 8/7/2013 until the last patient enrollment on 11/5/2015.
Description: The oversight total number of participants at risk was 200. Serious or non-serious adverse events were collected/assessed, but none observed.
Arm/Group | Dry Eye | Controls
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/33
Other Adverse Events (participants affected / at risk) | 0/167 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No